CLINICAL TRIAL: NCT00199953
Title: Post-nasal Drainage as an Extraesophageal Manifestation of Reflux
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Ortho-McNeil, Inc. (Industry); Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: RAB-USA-57; IRB numbers:; FMLH # 02-033; HRRC # 056-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2013-11

CONDITIONS: Postnasal Drainage
Keywords: Postnasal drainage; Extraesophageal reflux
MeSH Terms: interventions — Rabeprazole

INTERVENTIONS:
Drug: Rabeprazole 20 mg twice a day for 90-day period treatment

SUMMARY:
Objectives of this study are:

* To quantitatively evaluate the relationship between extraesophageal manifestations of gastroesophageal reflux (EER) and postnasal drainage(PND)in a group of patients without radiographic or endoscopic evidence of sinonasal inflammatory disease.
* To assess the efficacy of BID proton pump inhibitors (PPI) in the management of patients with symptomatic postnasal drainage.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease(GERD) is a common disorder of the esophagus, affecting 7-10% of the U.S. population. Characteristic symptoms include heartburn, chest pain, and indigestion. EER denotes gastroesophageal refluxate that reaches structures above the upper esophageal sphincter. EER has been implicated in the pathogenesis of several otolaryngologic disorders such as chronic posterior laryngitis, laryngeal contact ulcer or granuloma, paroxysmal laryngospasm, vocal cord nodules, Reinke's edema, subglottic or laryngotracheal stenosis, globus pharyngeus,and laryngeal and hypopharyngeal carcinoma. In addition, EER has been associated with disorders of both the lower and upper respiratory tract and with chronic sinonasal inflammation.

Patients with EER rarely complain of the common symptoms of GERD, such as heartburn. Often they present with symptoms involving the larynx and pharynx, including throat-clearing, globus pharyngeus, and postnasal drainage. These symptoms may be present due to direct irritation of the nasal epithelium by gastric refluxate and/or a neurogenic inflammatory process mediated by the autonomic nervous system.

Specific Aims:

* Specific Aim 1: To establish the relation ship between EER and PND in patients without sinonasal inflammatory disease.
* Hypothesis 1: In patients without radiographic or endoscopic evidence of sinonasal inflammatory disease, PND is a symptom of EER.
* Method 1: We will test this hypothesis utilizing a 2-site 24-hour pH probe test in a symptomatic patient group and compare then to a previously tested age and sex-matched control group.
* Specific Aim 2: To establish the efficacy of PPI in the management of PND.
* Hypothesis 2: Patients with a chief complaint of PND and no sinonasal inflammatory disease will improve with 3-month PPI treatment with Rabeprazole 20 mg twice a day.
* Method 2: A group of patients with a chief complaint of postnasal drainage, without radiographic or endoscopic evidence of sinonasal inflammatory disease will be entered into a prospective placebo-controlled trial utilizing BID PPIs over a 3-month period. the primary outcome measures will be: 1) Visual analog Scales, assessing the severity and frequency of PND at days 0 and 90 of treatment and 2)A quantitative color analysis of laryngeal erythema, utilizing videolaryngoscopy at days 0 and 90 of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and <70;
* PND as chief complaint;
* No known acute or chronic sinus disease;
* Nonsmokers;
* Subjects with no history of esophageal or gastric surgery
* Subjects with no history of allergic disease
* Women non pregnant.

Exclusion Criteria:

* Age , 18 or > 70;
* No PND as chief complaint
* Al;ergic disease or acute or chronic sinus disease;
* Smokers;
* Pregnant women;
* Subjects with history of esophageal or gastric surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
- VAS1:Visual Analog Scale indicating severity of PND
- VAS2:Visual Analog Scale indicating frequency of PND
- VAS3:Visual Analog Scale indicating frequency of throat-clearing.

SECONDARY OUTCOMES:
- Two-site 24-hour pH probe test indicating presence or gastroesophageal reflux episodes.
- Videolaryngoscopy for quantitative color analysis evaluation of laryngeal erythema as index of EER.

CONTACTS AND LOCATIONS:
Overall Officials: Todd A Loehrl, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Ulualp SO, Toohill RJ. Laryngopharyngeal reflux: state of the art diagnosis and treatment. Otolaryngol Clin North Am. 2000 Aug;33(4):785-802. doi: 10.1016/s0030-6665(05)70244-9. PMID 10918661
- [Background] Lodi U, Harding SM, Coghlan HC, Guzzo MR, Walker LH. Autonomic regulation in asthmatics with gastroesophageal reflux. Chest. 1997 Jan;111(1):65-70. doi: 10.1378/chest.111.1.65. PMID 8995994
- [Background] Chambers DW, Davis WE, Cook PR, Nishioka GJ, Rudman DT. Long-term outcome analysis of functional endoscopic sinus surgery: correlation of symptoms with endoscopic examination findings and potential prognostic variables. Laryngoscope. 1997 Apr;107(4):504-10. doi: 10.1097/00005537-199704000-00014. PMID 9111381
- [Background] Ulualp SO, Toohill RJ, Hoffmann R, Shaker R. Possible relationship of gastroesophagopharyngeal acid reflux with pathogenesis of chronic sinusitis. Am J Rhinol. 1999 May-Jun;13(3):197-202. doi: 10.2500/105065899781389777. PMID 10392238
- [Background] Jaradeh SS, Smith TL, Torrico L, Prieto TE, Loehrl TA, Darling RJ, Toohill RJ. Autonomic nervous system evaluation of patients with vasomotor rhinitis. Laryngoscope. 2000 Nov;110(11):1828-31. doi: 10.1097/00005537-200011000-00012. PMID 11081594
- [Background] Smit CF, Tan J, Devriese PP, Mathus-Vliegen LM, Brandsen M, Schouwenburg PF. Ambulatory pH measurements at the upper esophageal sphincter. Laryngoscope. 1998 Feb;108(2):299-302. doi: 10.1097/00005537-199802000-00027. No abstract available. PMID 9473087
- [Background] Hanson DG, Jiang J, Chi W. Quantitative color analysis of laryngeal erythema in chronic posterior laryngitis. J Voice. 1998 Mar;12(1):78-83. doi: 10.1016/s0892-1997(98)80077-5. PMID 9619981
- [Background] El-Serag HB, Lee P, Buchner A, Inadomi JM, Gavin M, McCarthy DM. Lansoprazole treatment of patients with chronic idiopathic laryngitis: a placebo-controlled trial. Am J Gastroenterol. 2001 Apr;96(4):979-83. doi: 10.1111/j.1572-0241.2001.03681.x. PMID 11316215
- [Background] Smith TL, Correa AJ, Kuo T, Reinisch L. Radiofrequency tissue ablation of the inferior turbinates using a thermocouple feedback electrode. Laryngoscope. 1999 Nov;109(11):1760-5. doi: 10.1097/00005537-199911000-00007. PMID 10569403